CLINICAL TRIAL: NCT02189421
Title: Comparison of Multibending and Conventional Ultra-slim Upper Endoscope for the Direct Advance Into the Bile Duct Without Assisting Accessory in Peroral Cholangioscopy
Brief Title: Multibending vs Conventional Endoscope for Direct Peroral Cholangioscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jong Choi, Assistant professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SCHBC 2014-06-012-001
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Common Bile Duct Calculi; Biliary Tract Cancer; Biliary Stricture; Bile Duct Diseases
Keywords: peroral cholangioscopy; ultra-slim upper endoscope; multibending endoscope
MeSH Terms: conditions — Gallstones; Biliary Tract Neoplasms; Bile Duct Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Direct peroral cholangioscopy (Other): Direct peroral cholangioscopy by using an ultra-slim upper endoscope without assisting accessories
  Interventions: Device: ultra-slim upper endoscope

INTERVENTIONS:
Device: ultra-slim upper endoscope — Direct peroral cholangioscopy by using an ultra-slim upper endoscope without assisting accessories
  Other Names: CHF-Y0009; GIF-XP290N

SUMMARY:
The aim of this study is to evaluate the usefulness of a newly developed multibending ultra-slim upper endoscope for the successful direct peroral cholangioscopy (POC) without assisting accessory in comparison with conventional ultra-slim endoscope. The investigators expect that multibending endoscope will show more higher successful performance than conventional endoscope.

DETAILED DESCRIPTION:
Direct POC using an ultra-slim upper endoscope permits various diagnostic and/or therapeutic intraductal interventions under direct endoscopic visualization in selected patients who has dilated distal CBD and widened papillary orifice. Because the bile duct has anatomical position in acute angle with the duodenum, assisting accessories such as intraductal anchoring balloon, guidewire or overtube is usually required for the successful direct POC. Recently, direct peroral cholangioscopes have been developed for free-hand direct advancement of the endoscope into the bile duct from duodenum. Multibending ultra-slim endoscope may be expected to facilitate the advance into the bile duct by overcoming the acute angle between the bile duct and the duodenum. After randomization of enrolled patients into two groups, direct POC will be performed by using a conventional slim endoscope in control group and by using a multibending endoscope in study group.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatobiliary diseases that are indicated for direct POC
* The patient who aged from 20 to 80 years. Legally acceptable representative must be capable of giving written informed consent prior to participation in this study
* The woman of child-bearing age must be negative from the pregnancy test in order to participate in this study
* Dilated common bile duct (> 8 mm)
* Having previous sphincterotomy and/or papillary balloon dilation
* The patients should not have any unacceptable conditions (e.g., physiological, familyish, social, geographical) for medical follow-up and adaptation of the study.

Exclusion Criteria:

* Contraindicated for ERCP
* Patients with stricture on papillary orifice
* Patients with periampullary malignancy
* Bleeding tendency: International normalized ratio (INR) of prothrombin time < 1.5 or platelet count < 60,000/mm3
* Patients with other serious disease or medical condition
* Patients with past medical history of significant neurologic or Psychiatric disorders such as dementia or seizure
* Unstable heart disease despite of treatment, recent myocardial infarction within 6 month (Even though MI was diagnosed within 6 months, if it becomes stable presently, the patient can be possible to participate).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Technical success of the direct peroral cholangioscopy | 6 months
  Successful insertion of a slim endoscope into the bile duct in no assisting accessories.

SECONDARY OUTCOMES:
Adverse events associated with direct POC | 6 months
  1. Cholangitis: fever and abdominal pain with abnormal liver function test
  2. Hemobilia: bleeding from the bile duct
  3. Pancreatitis: abdominal pain with elevation of the serum amylase and lipase
  4. Bile duct perforation: any evidence of bile duct perforation in imaging studies.
  5. Air embolism: clinical and imagine findings with air embolism

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Moon, MD, PhD, Principal Investigator — SoonChunHyang University School of Medicine
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, South Korea

REFERENCES:
- [Derived] Lee YN, Moon JH, Lee TH, Choi HJ, Itoi T, Beyna T, Neuhaus H. Prospective randomized trial of a new multibending versus conventional ultra-slim endoscope for peroral cholangioscopy without device or endoscope assistance (with video). Gastrointest Endosc. 2020 Jan;91(1):92-101. doi: 10.1016/j.gie.2019.08.007. Epub 2019 Aug 20. PMID 31442395